CLINICAL TRIAL: NCT03627403
Title: A Phase II Study to Evaluate the Efficacy and Safety of Selinexor in Patients With Myelofibrosis Refractory or Intolerant to JAK1/2 Inhibitors
Brief Title: Selinexor in Myelofibrosis Refractory or Intolerant to JAK1/2 Inhibitors
Acronym: ESSENTIAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI and Sponsor decision. Accrual was low and there was sufficient data to detect a response.
Sponsor: University of Utah (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI114354
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Primary Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Post-polycythemia Vera Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — selinexor

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized, prospective, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Selinexor, all patients (Experimental): Single Arm Study, all patients will get selinexor
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Selinexor will be administered orally at a dose of 80 mg once weekly until IWG-MR disease progression, intolerable toxicity, or no clinical benefit per treating physician's discretion whichever occurs first.
  For patients enrolled after Protocol v7, Selinexor will be administered by oral route beginning at 40mg once weekly. Prior to protocol version 7, the starting dose of sSelinexor was 60 mg and 80 mg once weekly.

SUMMARY:
This is a phase II, open label, prospective, single-arm study evaluating the efficacy and safety of selinexor in patients with PMF or secondary MF (PPV-MF or PET-MF) who are refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Diagnosis of primary myelofibrosis (PMF), post-essential thrombocytosis (PET-MF) or post-polycythemia vera (PPV-MF).
* Life expectancy ≥ 6 months.
* Prior treatment with ruxolitinib or any experimental JAK1/2 inhibitor with any one or more of the following:

  a. Inadequate response after being on ≥ 3 months of treatment defined by: i. Palpable spleen ≥ 10 cm below the left subcostal margin on physical examination at the screening visit OR ii. Palpable spleen ≥ 5cm below the left subcostal margin on physical examination at the screening visit AND active symptoms of MF at the screening visit defined presence of 1 symptom score of ≥ 5 or two symptom scores each of ≥ 3 using the Screening Symptoms Form (Appendix 6) b. Intolerant to ruxolitinib and/or other JAK1/2 inhibitors due to any grade ≥ 3 non-hematologic AEs of or any grade ≥ 2 AEs requiring treatment discontinuation AND palpable spleen ≥ 5cm below the left subcostal margin on physical examination at the screening visit.
* Adequate organ function as defined as:

  * Hematologic (≤ 28 days prior to C1D1):

    * Total white blood cell (WBC) count ≥ 1000/mm3
    * Absolute neutrophil count (ANC) ≥ 500/mm3
    * Hemoglobin ≥ 7 g/dL
    * Platelet count ≥ 30,000/mm3

For patients receiving transfusion and growth factor support, the following delays must be observed between the last administration and hematologic laboratory screening assessments:

• For hematopoietic growth factor support (including erythropoietin, darbepoetin, granulocyte-colony stimulating factor [G-CSF], granulocyte macrophage-colony stimulating factor [GM-CSF], and platelet stimulators [e.g., eltrombopag, romiplostim, or interleukin-11]): at least 2 weeks.

Growth factor support, RBC and/or platelet transfusions are allowed as clinically indicated per institutional guidelines during the study.

* Hepatic (≤ 28 days prior to C1D1):

  * Total bilirubin < 1.5 × ULN except in patients with indirect hyperbilirubinemia due to hemolysis or with Gilbert's syndrome where total bilirubin should be < 5 × ULN
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 × ULN.
* Renal (within 28 days prior to C1D1):

  * Estimated creatinine clearance (CrCl) ≥ 20 mL/min using the Cockcroft and Gault formula [(140-Age) × Mass (kg)/(72 × creatinine mg/dL), multiply by 0.85 if the patient is female] OR

    * Female patients of childbearing potential must have a negative serum pregnancy test (≤ 3 days prior to C1D1).
    * Female patients of childbearing potential must agree to use 2 methods of contraception throughout the study and for 3 months following the last dose of study treatment (including 1 highly effective and 1 effective method of contraception as defined in section 7.4)
    * Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential.
    * Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior treatments including ruxolitinib or other experimental agents unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
    * Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior exposure to a SINE compound, including selinexor.
* Patients who are below their ideal body weight and would be unduly impacted by changes in their weight, in the opinion of the investigator, will be excluded
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals ≤ 1 week prior to C1D1. Patients on prophylactic antibiotics or with a controlled infection ≤ 1 week prior to C1D1 are acceptable.
* Radiation, chemotherapy, immunotherapy, or any other anticancer therapy (including investigational therapies) ≤ 2 weeks.
* Ruxolitinib or other JAK1/2 inhibitors ≤ at least 3 days or 5 half-lives prior to C1D1.
* Major surgery ≤ 4 weeks prior to C1D1.
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus ribonucleic acid (RNA) or hepatitis B virus surface antigen.
* Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
* Any life-threatening illness, organ system dysfunction, or serious psychiatric, medical, or other conditions/situations which, in the investigator's opinion, could compromise a patient's ability to give informed consent, safety, or compliance with the protocol.
* Contraindication to any of the required concomitant drugs or supportive treatments.
* Subjects taking prohibited medications as described in Section 6.3. Following discontinuation of prohibited medications, a washout period is required prior to initiating study treatment (the duration of the washout must be as clinically indicated, e.g. at least five half-lives).
* Subjects who are breastfeeding and unwilling to stop while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2025-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Tantravahi, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor, All Patients: Single Arm Study, all patients received selinexor.
  Selinexor: Selinexor was administered weekly until IWG-MR disease progression, intolerable toxicity, or no clinical benefit per treating physician's discretion whichever occurs first.
  For patients enrolled after Protocol v7, Selinexor was administered by oral route beginning at 40mg once weekly. Prior to protocol version 7, the starting dose of Selinexor was 60 mg and 80 mg once weekly.
Period: Overall Study
Arm/Group | Selinexor, All Patients
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selinexor, All Patients
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.82 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Diagnosis [Count of Participants; unit: Participants]
  Primary Myelofibrosis (PMF) | 8
  Post-Essential Thrombocytosis (PET-MF) | 4
  Post-Polycythemia Vera (PPV-MF) | 5
Hemoglobin [Count of Participants; unit: Participants]
  >= 10 g/dL | 8
  < 10 g/dL | 9
WBC [Count of Participants; unit: Participants]
  <= 25 cells x 10^9/L ( <= 25 k/uL) | 17
  > 25 cells x 10^9/L) ( > 25 k/uL) | 0
Peripheral blood blast [Count of Participants; unit: Participants] — Peripheral blood blasts are immature white blood cells, and their presence can indicate a blood disorder or cancer. Several prognostic scoring systems have been developed for Myelofibrosis and are currently used in the clinic to estimate survival, risk of leukemic transformation, and also guide treatment decisions. One such system, International Prognostic Scoring System (IPSS), was developed based on certain clinical features at diagnosis including peripheral blood blasts > 1% among other factors.
  Participants
    < 1 % | 8
    >= 1 % | 9
Constitutional symptoms [Count of Participants; unit: Participants] — Constitutional symptoms include weight loss>10% of the baseline value in the year preceding Primary Myelofibrosis (PMF) diagnosis and unexplained fever or excessive sweats persisting for more than one month. Constitutional symptoms are one of the five variables scored on the Primary Myelofibrosis Dynamic International Prognostic Scoring System (DIPSS), which is used to predict survival and risk in patients with PMF.
  Participants
    Yes | 7
    No | 10
DIPSS Risk Group [Count of Participants; unit: Participants] — The Dynamic International Prognostic Scoring System (DIPSS) risk assessment is used to predict overall survival (OS) and risk in patients with PMF. It consists of five variables: Age > 65 years (1 pt), Hemoglobin < 10 g/dL (2 pts), White Blood Cells > 25 K/uL (1 pt), Circulating Blasts ≥ 1% (1 pt), and Constitutional Symptoms (1 pt).
  DIPSS Risk Groups are based on the total points. The groups are Low Risk (0 pts; median OS not reached), Intermediate-1 (1 to 2 pts; median OS 14.2 years), Intermediate-2 (3 to 4 pts; median OS 4 years), and High (5 to 6 pts; median OS 1.5 years).
  Participants
    Low | 1
    Intermediate-1 (INT-1) | 7
    Intermediate-2 (INT-2) | 9
    High | 0
Weight [Mean (Standard Deviation); unit: kg] | 85.17 (19.13)
Height [Mean (Standard Deviation); unit: cm] | 173.19 (11.17)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.36 (5.79)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Reduction in Spleen Volume
Description: To assess the efficacy of selinexor on spleen volume reduction in subjects with myelofibrosis (PMF, PET-MF, or PPV-MF) refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.
  This outcome will report the number of subjects with ≥ 35% reduction in spleen volume as measured by MRI or CT abdomen from baseline to after six cycles of treatment or end of treatment. Patients who did not complete six cycles of treatment received an MRI at discontinuation of therapy. Patients who died prior to completing six cycles of treatment or a follow-up scan were considered non-responders.
Time Frame: Up to 5.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, All Patients
Number analyzed (Participants) | 17
Participants | 3

2. Secondary Outcome: Adverse Events That Occur
Description: To assess the safety/tolerability and further characterize the safety profile of selinexor in PMF, PET-MF, or PPV-MF patients refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.
  Secondary Endpoints: rate of adverse events (AEs) and serious adverse events (SAEs).
Time Frame: Up to 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Percent Change of Spleen Volume
Description: To further assess the efficacy and clinical activity of selinexor (by means of overall response) in subjects with myelofibrosis (PMF, PET-MF, or PPV-MF) refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.
  This outcome will report the mean percent change of spleen volume as measured by MRI or CT abdomen from baseline to after six cycles of treatment or end of treatment. Patients who did not complete six cycles of treatment received an MRI at discontinuation of therapy. Patients who died prior to completing six cycles of treatment or a follow-up scan were not included in this endpoint.
  The mean and standard will be reported for the change in spleen volume.
Time Frame: Up to 5.5 months
Population: One participant did not reach this endpoint. This participant only completed a baseline disease assessment.
Measure: Mean (Standard Deviation); unit: percent (%) change of spleen volume
Arm/Group | Selinexor, All Patients
Number analyzed (Participants) | 16
percent (%) change of spleen volume | 2.96 (37.64)

4. Secondary Outcome: Change in Symptoms Score
Description: To further assess the efficacy and clinical activity of selinexor (by means of reduction in symptoms) in subjects with myelofibrosis (PMF, PET-MF, or PPV-MF) refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.
  This outcome reports the count of patients with ≥ 50% reduction of total symptoms scores as measured by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) from baseline after 6 cycles of treatment. Patients who did not complete 6 cycles of treatment will receive the MPN-SAF assessment at discontinuation of therapy.
  The MPN-SAF is a symptom assessment completed by the patients including fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the sum of all the individual scores (0-100 scale).
Time Frame: Up to 5.5 months
Population: One participant was not evaluable for this endpoint; this participant did not complete a baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor, All Patients
Number analyzed (Participants) | 16
Participants
  ≥ 50% Reduction of MPN-SAF TSS Score | 2
  < 50% Reduction of MPN-SAF TSS Score | 14

5. Secondary Outcome: Overall Response
Description: To further assess the efficacy and clinical activity of selinexor (by means of overall response) in subjects with myelofibrosis (PMF, PET-MF, or PPV-MF) refractory or intolerant to ruxolitinib and/or any other experimental JAK1/2 inhibitors.
  Overall response according to the 2013 International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) consensus criteria for treatment response in primary and secondary MF (post-PV and post-ET). The IWG-MRT response categories are CR (Complete Response), PR (Partial Response), CI (Clinical Improvement), Anemia Response, Spleen Response, Symptoms Response, Progressive Disease, Stable Disease, Relapse.
Time Frame: Up to 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: Overall survival at 24 months from the initiation of study therapy.
Time Frame: Up to 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the first dose of study until end of treatment (up to 16.6 months). Currently three subjects are still on treatment and adverse event collection is still ongoing.
Groups:
- Selinexor, All Patients: Single Arm Study, all patients received selinexor.
  Selinexor: Selinexor was administered weekly until IWG-MR disease progression, intolerable toxicity, or no clinical benefit per treating physician's discretion whichever occurs first.
  For patients enrolled after Protocol v7, Selinexor was administered by oral route beginning at 40mg once weekly. Prior to protocol version 7, the starting dose of Selinexor was 60 mg and 80 mg once weekly.
  Participants experienced dose escalations and reductions based on their individual responses. Subjects were not assigned to fixed-dosing cohorts as dosing ranged from 20mg once weekly to 80 mg once weekly. Adverse Events were not collected specific to dose.
Arm/Group | Selinexor, All Patients
All-Cause Mortality (participants affected / at risk) | 6/17
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor, All Patients (N=17)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor, All Patients (N=17)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (21)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Anorexia (Metabolism and nutrition disorders) | 11 (13)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Belching (Gastrointestinal disorders) | 1 (3)
Bloating (Gastrointestinal disorders) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (3)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cataract (Eye disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (14)
Dizziness (Nervous system disorders) | 7 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 8 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 5 (10)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 12 (22)
Fever (General disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (4)
Flu like symptoms (General disorders) | 3 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (4)
Gum infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (8)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Malaise (General disorders) | 1 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 15 (20)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Periorbital edema (Eye disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (8)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Testosterone deficiency (Endocrine disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 7 (9)
Weight loss (Investigations) | 8 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03627403/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03627403/ICF_001.pdf